CLINICAL TRIAL: NCT00336427
Title: A Prospective Study of MRSA Colonization in Peripartum Women and Their Offspring
Brief Title: MRSA Colonization in Peripartum Women and Their Offspring
Status: Completed | Type: Observational
Sponsor: Orlando Regional Medical Center (Other)
Collaborators: Pfizer (Industry)
Other Study IDs: ORMC-MRSA-Pregnancy
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Last update posted 2006-06-13 (Estimated); Status verified 2006-05

CONDITIONS: Pregnancy; Bacterial Colonization
Keywords: MRSA; Colonization; Pregnancy; Neonates

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
We hypothesize that pregnant women are at baseline risk for carrying community-acquired MRSA, but also have frequent contact with healthcare workers which may put them at risk for hospital-acquired MRSA carriage. Our study aimed to identify the colonization rate of women in active labor and whether transmission to infants may occur.

DETAILED DESCRIPTION:
Mothers are at risk for carrying MRSA. What this risk is is not known. We have seen a dramatic increase in neonatal intensive care unit MRSA infections. Could mothers transmit MRSA to their newborns if they are asymptomatic carriers? Mothers come into close contact with health care providers, often have other children in daycare (known risk factor) and may have other exposures to MRSA. Our study was designed to sample 300 mother-infant pairs to determine whether MRSA carriage is present in asymptomatic women. The study consisted of obtaining informed consent, then performing a sterile swab of mothers' nares and vaginal area, then babies' nares and umbilicus once the baby was born.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy expected to deliver next 24 hours

Exclusion Criteria:

* Cesarean sections

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2005-09; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Margret G Reusch, MD, Principal Investigator — ORMC